CLINICAL TRIAL: NCT06512090
Title: To Investigate the Effects of Low Glycemic Index（LGI）Related Steamed Bread on Glycemia Control, Islet Function in Patients With Type 2 Diabetes in China: A Single-center, Randomized, Open-label, Prospective Study
Brief Title: Effects of LGI Steam Bread on Glycemia Control in T2DM in China
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai Punan Hospital of Pudong New District (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2024009
Record Dates: First submitted 2024-07-16; First posted 2024-07-22 (Actual); Last update posted 2024-07-22 (Actual); Status verified 2024-07

CONDITIONS: Diabete Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Diet, Diabetic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- LGI steam bread intervention group (Experimental): The participant in this group takes LGI steam bread as staple food instead of diabetic diet during the study period.
  Interventions: Dietary Supplement: LGI steam bread
- Diabetic diet group (Active Comparator): he participant in this group takes diabetic diet during the study period.
  Interventions: Dietary Supplement: Diabetic diet

INTERVENTIONS:
Dietary Supplement: LGI steam bread — LGI Steam bread called "Mangu"steam bread
  Arms: LGI steam bread intervention group
Dietary Supplement: Diabetic diet — the calorie intake of Diabetic diet will by recommended by nutritionist
  Arms: Diabetic diet group

SUMMARY:
This was a single-center, randomized, open, prospective, parallel-controlled, head-to-head comparison trial. To investigate the effects of low glycemic index（LGI）related steam bread on glycemic control，islet function in patients with type 2 diabetes.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18yrs；
* Diagnosed as Type 2 Diabetes;
* Had been on a stable hypoglycemic regimen for at least 30 days prior to screening；
* HbA1c between 7.5% and 11.0% (both upper and lower limits included) in the 90 days prior to screening;
* Fasting C-peptide ≥1.0ng/ml in the 90 days prior to screening;
* Be willing to accept and adhere to LGI steamed bread as a staple food for at least 14 days

Exclusion Criteria:

* Diagnosed with type 1 diabetes, or secondary diabetes;
* Have clinically significant liver disease, moderate/severe kidney injury, or end-stage renal disease;
* Has unstable CV disorders, including heart failure (NYHA) class III or IV), intractable angina, uncontrolled arrhythmias, and severe uncontrolled hypertension (systolic blood pressure ≥180mmHg, or diastolic blood pressure ≥105mmHg);
* An Acute Coronary Syndrome event (ACS) occurred within the 6 months prior to randomization

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 144 (Estimated)
Dates: Start 2024-07-13 (Estimated); Primary Completion 2025-01-27 (Estimated); Study Completion 2025-02-28 (Estimated)

PRIMARY OUTCOMES:
glucose at 120 mins | 120 minutes
  the blood glucose level at 120 mins after Standard meal test

SECONDARY OUTCOMES:
glucose at 60 mins | 60 minutes
  The blood glucose at 60 mins after standard meal test
iAUC 120 minutes | 120 minutes
  120-minute Area under the Curve (iAUC)

CONTACTS AND LOCATIONS:
Overall Officials: LianYong Liu, ph.D, Principal Investigator — Shanghai Punan Hospital of Pudong New District

IPD SHARING:
Plan to Share IPD: No